Title of the study: Comparative effects of Kinesiotaping versus Pressure garments on secondary

upper extremity lymphedema following microsurgical breast reconstruction after severe chest

burns.

Date: 23/12/2023

Statistical analysis:

Subjects' personal and anthropometric measurements were calculated using Kolmogorov-

Smirnov test for testing homogeneity and the data were represented in tabular form. The

measurements were taken before the intervention, during the intervention, after at 4 weeks and 8

weeks after intervention and after 6 months follow up. The data were shown as mean and standard

deviation with a 95% confidence interval (CI) with an upper and lower limit. The time and group

(4 × 2) mixed model for repeated measures (MMRM) of primary and secondary variables are

reported between group A and group B at various intervals. Student's t-test was used to calculate

inter-group effects and repeated measures (rANOVA) were used to calculate the intra-group effects.

IBMSPSS – online version 20 was used to do all the statistical tests and the  $\alpha$  level was set at 0.05.